CLINICAL TRIAL: NCT02448862
Title: Differences in Incidence of Common Side Effects Between Young Adults and Elderly Patients While Using Fentanyl-based IV-PCA
Brief Title: Differences in Incidence of Common Side Effects Between Young Adults and Elderly Patients While Using IV-PCA
Status: Completed | Type: Observational
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Dr. Koh, Jae Chul, MD, Department of anesthesiology and pain medicine, Severance Hospital
Other Study IDs: 2015-0098-001
Record Dates: First submitted 2015-05-14; First posted 2015-05-20 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting
Keywords: IV-PCA; Elderly patients; Yound adults; Side effect; Postoperative pain; Postoperative nausea and vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Elderly patients: Patients aged over 70 who had used fentanyl based IV-PCA for postoperative pain.
  Interventions: Device: Fentanyl based IV-PCA
- Young adults: Patients aged 20 to 39 who had used fentanyl based IV-PCA for postoperative pain.
  Interventions: Device: Fentanyl based IV-PCA

INTERVENTIONS:
Device: Fentanyl based IV-PCA — We have used a disposable PCA pump (Ambix Anaplus®; E-Wha Fresenius Kabi, Korea or accufuser plus®; Woo Young Medical, Korea) and fentanyl was diluted in 100 mL with saline for 48 hrs PCA infusion. The pump was set as follows: infusion rate as 2 ml/hr, bolus dose as 0.5 ml or 1 ml, lockout time as 15 min. It was decided at the anesthesiologist's option whether the additional analgesic drug (ketorolac or nefopam) and the antiemetic drug (ondansetron, ramosetron or palonosetron) would be added in PCA or not. The anesthesiologist who performed the anesthesia decided the amount of chosen drugs.
  Other Names: Intravenous patient controlled analgesic device

SUMMARY:
In this retrospective study, postoperative pain score, PCA-related complications, the risk factors for requirement of rescue analgesics and antiemetics will be evaluated in young and elderly patients, respectively, using fentanyl-based IV PCA during postoperative 48 hours after various surgeries.

DETAILED DESCRIPTION:
Since 2010, A PCA service team in the investigators' hospital have collected multidisciplinary clinical data from all the patients who used IV-PCA postoperatively in aim of the assessment of clinical outcome. The investigators reviewed the collected data from the patients who had used IV-PCA for pain control after an elective surgery under general or spinal anesthesia between Sep. 2010 and March. 2014. The need for informed consent was waived for this study. The investigators have used a disposable PCA pump (Ambix Anaplus®; E-Wha Fresenius Kabi, Korea or accufuser plus®; Woo Young Medical, Korea) and fentanyl was diluted in 100mL with saline for 48 hrs PCA infusion. The pump was set as follows: infusion rate as 2 ml/hr, bolus dose as 0.5 ml or 1 ml, lockout time as 15 min. It was decided at the anesthesiologist's option whether the additional analgesic drug (ketorolac or nefopam) and the antiemetic drug (ondansetron, ramosetron or palonosetron) would be added in PCA or not. The anesthesiologist who performed the anesthesia decided the amount of chosen drugs. Exclusion criteria were as following: age < 20 years old, age 40 to 69, postoperative ventilator support or intensive care, and imperfect data. The data of the PCA regimen which has been decided were recorded and analyzed. Demographic variables including age, sex, body mass index, American Society of Anesthesiologists (ASA) physical status and history of smoking, motion sickness, postoperative nausea/vomiting, hypertension and diabetes mellitus have been analyzed. Anesthesia and surgery-related variables including the duration of anesthesia, the type of anesthesia (general or spinal), laparoscopy and the operation site (categorized in abdominal, thoracic, upper & lower extremities, head & neck, spine and others) were also been analyzed. PCA-related variables included total dose of fentanyl for two days (µg/kg), use of mixed additional analgesics and antiemetics in PCA and discontinuation of PCA. When the patient requested the discontinuation of IV-PCA, the reason and the time have been recorded. Postoperative variables including the numeric rating scale (NRS, 0-10, 0 = no symptom; 10= unthinkable worst pain) for pain, requirements of rescue analgesics and antiemetics were analyzed. And the postoperative complications including nausea, vomiting, headache, dizziness, and sedation were analyzed. All the postoperative variables were recorded at postoperative 0-6 hrs including stay at post-anesthesia care unit, 6-12, 12-18, 18-24 and 24-48 hrs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had used IV-PCA for pain control after an elective surgery under general or spinal anesthesia between Sep. 2010 and March. 2014

Exclusion Criteria:

* Age < 20 years old,
* age 40 to 69,
* postoperative ventilator support or intensive care,
* and imperfect data

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collected data from the patients who had used IV-PCA for pain control after an elective surgery under general or spinal anesthesia between Sep. 2010 and March. 2014.
Sampling Method: Non-Probability Sample
Enrollment: 10575 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Chul Koh, MD, Principal Investigator — Gang Nam Severance Hospitial
Locations (1):
- Gangnam Severance hospital, Seoul, Gangnam-gu, South Korea

REFERENCES:
- [Background] Choi JB, Shim YH, Lee YW, Lee JS, Choi JR, Chang CH. Incidence and risk factors of postoperative nausea and vomiting in patients with fentanyl-based intravenous patient-controlled analgesia and single antiemetic prophylaxis. Yonsei Med J. 2014 Sep;55(5):1430-5. doi: 10.3349/ymj.2014.55.5.1430. PMID 25048507
- [Background] Mortimer M, Ahlberg G; MUSIC-Norrtalje Study Group. To seek or not to seek? Care-seeking behaviour among people with low-back pain. Scand J Public Health. 2003;31(3):194-203. doi: 10.1080/14034940210134086. PMID 12850973

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elderly Patients | Young Adults
Started | 4525 | 6050
Completed | 4525 | 6050
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderly Patients | Young Adults | Total
Number analyzed (Participants) | 4525 | 6050 | 10575
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 6050 | 6050
  >=65 years | 4525 | 0 | 4525
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (4.4) | 31.7 (5.8) | 57.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2169 | 3706 | 5875
  Male | 2356 | 2344 | 4700
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 4525 | 6050 | 10575

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Rescue Analgesics Requirement
Description: The percentage of patients who required rescue analgesics at least once during the postoperative 48-hour period
Time Frame: Postoperative 48 hours
Measure: Number; unit: Percentage of Participants
Arm/Group | Elderly Patients | Young Adults
Number analyzed (Participants) | 4525 | 6050
Percentage of Participants | 47.9 | 53.8

2. Primary Outcome: Incidence of Rescue Antiemetics Requirement
Description: The proportion of patients who required rescue antiemetics at least once during the postoperative 48-hour period
Time Frame: Postoperative 48 hours
Measure: Number; unit: Percentage of Participants
Arm/Group | Elderly Patients | Young Adults
Number analyzed (Participants) | 4525 | 6050
Percentage of Participants | 12.2 | 10.1

3. Secondary Outcome: Postoperative Pain in Numeric Pain Scale
Description: The Numeric Pain Scale (NRS - 0: no pain, 10: worst pain can't imagine) for pain measured once at each time periods (0~6, 6~12, 12~18, 18~24, 24~48 hours)
Time Frame: Postoperative 48 hours
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elderly Patients | Young Adults
Number analyzed (Participants) | 4525 | 6050
Scores on a scale
  Postoperative 0-6 hours | 5.74 (1.90) | 5.70 (1.94)
  Postoperative 6-12 hours | 4.58 (1.8) | 4.68 (1.79)
  Postoperative 12-18 hours | 3.97 (1.63) | 3.91 (1.59)
  Postoperative 18-24 hours | 3.32 (1.46) | 3.33 (1.45)
  Postoperative 24-48 hours | 2.84 (1.32) | 2.83 (1.31)

4. Secondary Outcome: Incidence of Nausea and Vomiting
Description: The percentage of participants who had nausea and vomiting during postoperative 48 hours
Time Frame: Postoperative 48 hours
Measure: Number; unit: percentage of participants
Arm/Group | Elderly Patients | Young Adults
Number analyzed (Participants) | 4525 | 6050
percentage of participants | 20.6 | 23.8

5. Secondary Outcome: Incidence of Dizziness or Headaches
Description: The percentage of participants who had headache and dizziness
Time Frame: Postoperative 48 hours
Measure: Number; unit: percentage of participants
Arm/Group | Elderly Patients | Young Adults
Number analyzed (Participants) | 4525 | 6050
percentage of participants
  headache | 1.7 | 2.3
  dizziness | 6.5 | 9.8

ADVERSE EVENTS:
Arm/Group | Elderly Patients | Young Adults
Serious Adverse Events (participants affected / at risk) | 0/4525 | 0/6050
Other Adverse Events (participants affected / at risk) | 0/4525 | 0/6050

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No